CLINICAL TRIAL: NCT02133417
Title: A Prospective Multi-center Case Collection Study of Breast Imaging Examinations From Women With Mammographically-detected Lesion(s) to Evaluate the Non-inferiority of Digital Mammography (XRM) and Quantitative Transmission Ultrasound (QTUS) Together Compared to XRM and Hand Held Ultrasound (HHUS) Together in the Evaluation of Lesion(s) Detected With Diagnostic Mammography.
Brief Title: Non-Inferiority Quantitative Transmission Ultrasound Case Collection Study
Acronym: QTUS
Status: Completed | Type: Observational
Sponsor: QT Ultrasound LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013001
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Mass Lesion
Keywords: Quantitative Transmission Ultrasound; QTUS

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women: Women with mammographically-detected breast lesions
  Interventions: Device: Quantitative Transmission Ultrasound

INTERVENTIONS:
Device: Quantitative Transmission Ultrasound — Quantitative Transmission Ultrasound (QTUS) as an automated breast ultrasound procedure for women who have a mammographically detected mass.
  Other Names: QTUS; QT Ultrasound

SUMMARY:
Conduct a case collection study of breast imaging examinations from women with mammographically-detected breast lesions for the purpose of conducting subsequent Reader Studies.

DETAILED DESCRIPTION:
This is a prospective case collection study for the purpose of collecting cases for the subsequent Reader Studies at a minimum of two clinical sites.

Potential subjects will be recruited from a group of women who have undergone diagnostic mammography and demonstrate a mammographic lesion in at least one view. Approximately 300 women will be enrolled. Subjects will undergo QTUS following a diagnostic XRM with a mammographically-detected lesion(s) in at least one mammographic view and will have a lesion seen on HHUS corresponding to the XRM lesion(s). Potential Subjects will be eligible for enrollment at the time the corresponding lesion is identified on HHUS. All subjects will undergo an ultrasound guided aspiration/biopsy with cytology to determine whether the lesion is a cyst or solid.

Each study site is projected to collect approximately 75 cyst cases and 75 solid cases for a total of 150 cases, stratified across the four (4) recognized breast tissue density categories with at least 50% of cases from subjects with heterogeneous and extremely dense breast compositions. The composition of the cyst cases at each site is projected to consist of 25 simple cysts and 50 complicated and complex cysts for a total of 75 cyst cases. All enrolled subjects will undergo ultrasound guided aspiration or biopsy or surgical excision, as applicable for the index lesion. Cytologic or histologic results for all lesions will be performed and collected.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 25 or older
* A bra cup size of A through DDD
* Willing and able to provide written, signed Informed Consent Form (ICF) after the nature of the study has been explained, all questions have been answered, and prior to any research-related procedure(s)
* Willing and able to comply with all study procedure(s), including possible aspiration for a simple cyst
* Complete digital mammography views Craniocaudal and Medio-lateral Oblique (CC and MLO) for one or both breasts
* Mammographically-detected lesion(s) seen on at least one mammographic view and a corresponding HHUS correlate(s)

Exclusion Criteria:

* Does not meet all Inclusion Criteria
* Currently breastfeeding
* History of breast cancer in the past 12 months, except for Fine Needle Aspirations (FNA) or Cyst Aspiration
* History of breast surgeries or interventional breast procedures in the past 12 months
* Normal mammogram at the time of this evaluation
* Physical inability to tolerate the procedure on the scanner, i.e. inability to lie prone and still for up to 30 minutes at a time
* Open wounds, sores or skin rash present on the breast(s) or nipple discharge from the scanned breast
* Breasts too large for scanner, i.e. bra size larger than DDD or inability to successfully "fit" breast after the subject is placed on scanner
* Body weight greater than 400 lbs. (180 kg)
* Has a concurrent disease or condition which in the judgment of the principal investigator disqualifies the subject, from participating in the study

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligibility for enrollment will be open to women of all races and ethnicities who have completed a diagnostic XRM with a mammographically-detected lesion(s) in at least one mammographic view and have a lesion seen on HHUS corresponding to the XRM lesion(s). Women with a normal mammogram at the time of this evaluation are not eligible to participate. Women younger than 25 years of age will not be eligible to participate. Potential subjects must not be breastfeeding at the time of diagnostic breast imaging. Patients who have had breast cancer, breast surgeries, or interventional breast procedures in the past 12 months will not be eligible to enter the study.
Sampling Method: Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The purpose of the case collection study is to collect mammographically-detected breast lesions seen in at least one mammographic view in the clinical setting and seen on HHUS, and confirmed by pathology. | 12 months
  This is a prospective Case Collection study for the purpose of conducting subsequent Reader Studies. The primary objective for this prospective case collection study is to provide up to 300 cytology/pathology confirmed cases for subsequent Reader Studies.

CONTACTS AND LOCATIONS:
Overall Officials: Rajni Natesan, MD, Study Director — Chief Medical Officer
Locations (2):
- United States (2):
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Elizabeth Wende Breast Care, LLC, Rochester, New York